CLINICAL TRIAL: NCT03460522
Title: Open Label Phase II Study to Evaluate the Efficacy and Safety of Inotuzumab Ozogamicin for Induction Followed by Chemotherapy Consolidation and Maintenance Therapy In Patients Aged 56 Years and Older With Acute Lymphoblastic Leukemia (ALL)
Brief Title: Inotuzumab Ozogamicin and Conventional Chemotherapy In Patients Aged 56 Years and Older With ALL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nicola Goekbuget (Other)
Responsible Party: Sponsor-Investigator, Nicola Goekbuget, Head of GMALL, Goethe University
Organization: Goethe University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INITIAL-1
Record Dates: First submitted 2018-02-22; First posted 2018-03-09 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Precursor Cell Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction Therapy with Inotuzumab Ozogamicin (Experimental): Patients will receive up to 3 cycles Inotuzumab with applications on day 1, 8 and 15 in each cycle. First dose will be 0.8 mg/m² on Day 1. All subsequent doses will be 0,5 mg/m².
  Interventions: Drug: Inotuzumab ozogamicin

INTERVENTIONS:
Drug: Inotuzumab ozogamicin — Patients will receive standard of care chemotherapy (only maintenance) after Inotuzumab Ozogamicin.

SUMMARY:
The trial proposed to evaluate the efficacy and safety of an inotuzumab ozogamicin followed by maintenance treatment in patients with acute lymphoblastic leukemia older than 56 years

DETAILED DESCRIPTION:
Despite recent advances especially in younger patients, the prognosis of elderly patients with ALL remains dismal with a 5-year survival rate of around 20%, even after intensive chemotherapy.

Inotuzumab ozogamicin (PF-05208773; CMC-544) is an antibody-targeted intravenous (IV) chemotherapy agent composed of an anti-CD22 antibody linked to calicheamicin, a potent cytotoxic antitumor antibiotic.

After a prephase treatment, induction therapy will be based on three cycles of inotuzumab ozogamicin and intrathecal therapy only. This will be followed by a conventional maintenance therapy. All patients will be followed for cytological response, minimal residual disease and safety parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ≥56 years of age and contraindication for age-adapted consolidation chemotherapy due to age (≥75 years) and/or severe co-morbidities (>2 per Charlson Score).
2. Newly diagnosed acute lymphoblastic leukemia (>25% marrow blasts, assessed by morphology; i.e. M3 marrow)
3. Leukemic blasts must have CD22 surface expression of at least 20%, assessed by local/institutional flow cytometry of a bone marrow aspirate sample (assessment of CD22 via the reference lab for immunophenotyping is strongly recommended). In the case of an inadequate aspirate sample (dry tap), flow cytometry of peripheral blood specimen may be substituted if the patient has circulating blasts; alternatively, CD22 expression may be documented by immunohistochemistry of a bone marrow biopsy specimen
4. No previous ALL-specific treatment with the exception of corticosteroids and/or single dose vincristine and/or a maximum of three doses of cyclophosphamide (cumulative dose of 600 mg/m2) and the standard prephase treatment
5. With or without documented CNS involvement
6. Adequate liver function, including total serum bilirubin < 2.0 x upper limit of normal (ULN) unless the patient has documented Gilbert syndrome, and aspartate and alanine aminotransferase (AST and ALT) < 2.5 x ULN. If organ function abnormalities are considered due to leukemic infiltration of the liver, total serum bilirubin must be < 2.5 x ULN and AST/ALT < 5 x ULN
7. Serum creatinine <1.5 x ULN or any serum creatinine level associated with a measured or calculated creatinine clearance of >40 mL/min
8. WHO performance status ≤ 2
9. Signed written inform consent
10. Inclusion in GMALL registry

Exclusion Criteria:

1. Philadelphia-chromosome or BCR-ABL positive ALL
2. Burkitt's or mixed phenotype acute leukemia based on the WHO 2008 criteria
3. Peripheral absolute lymphoblast count >10,000/μL after pre-phase treatment and before start of study medication
4. Known systemic vasculitis (e.g. , Wegener's granulomatosis, polyarteritis nodosa, systemic lupus erythematosus), primary or secondary immunodeficiency (such as HIV infection or severe inflammatory disease)
5. Current or chronic hepatitis B or C infection as evidenced by hepatitis B surface antigen and anti-hepatitis C antibody positivity, respectively, or known seropositivity for human immunodeficiency virus (HIV)
6. Major surgery within < 4 weeks before entry on study
7. Unstable or severe uncontrolled medical condition (e.g., unstable cardiac function or unstable pulmonary condition)
8. Concurrent active malignancy other than non-melanoma skin cancer, carcinoma in situ of the cervix, or localized prostate cancer that has been definitely treated with radiation or surgery; patients with previous malignancies are eligible provided that they have been disease free for >2 years
9. Cardiac function, as measured by left ventricular ejection fraction (LVEF) that is less than 45%, or the presence of New York Heart Association (NYHA) stage III or IV congestive heart failure
10. Myocardial infarction < 6 months before entry on study
11. History of clinically significant ventricular arrhythmia, or unexplained syncope not believed to be vasovagal in nature, or chronic bradycardic states such as sinoatrial block or higher degrees of AV block unless a permanent pacemaker has been implanted
12. Uncontrolled electrolyte disorders that can confound the effects of a QTc prolonging drug (e.g., hypokalemia, hypocalcemia, hypomagnesemia)
13. History of chronic liver disease (e.g., cirrhosis) or suspected alcohol abuse
14. History of hepatic veno-occlusive disease (VOD) or sinusoidal obstruction syndrome (SOS)
15. Administration of live vaccine <6 weeks before entry on study
16. Evidence of uncontrolled current serious active infection (including sepsis, bacteremia, fungemia or COVID-19 infection) or patients with a recent history (within 4 months) of deep tissue infections such as fasciitis or osteomyelitis
17. Patients who have had a severe allergic reaction or anaphylactic reaction to any humanized monoclonal antibodies or any known hypersensitivity to the active substance or any of its excipients
18. Pregnant females; breastfeeding females; males and females of childbearing potential (a woman is considered of childbearing potential (WOCBP) i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile e.g. after hysterectomy or bilateral ovariectomy. Please refer to chapter 12.4 Contraceptive Requirements.) not using highly effective contraception or not agreeing to continue highly effective contraception for women at least 8 months and for men at least 5 months after the last dose of investigational product

18. Participation in other studies involving investigational drug(s) (Phase I-IV) within 4 weeks before study inclusion

19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Ages: 56 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) at 12-months follow-up | At 12 months
  An event is any of the following: persisting bone marrow blasts (more than 5% leukemic blasts) after two cycles of inotuzumab ozogamicin, relapse or death.

SECONDARY OUTCOMES:
Complete hematological remission | 42 days
  The rate of complete hematological remission after inotuzumab ozogamicin induction treatment
MRD response after induction treatment | 42 days
  The rate of patients being negative for minimal residual disease (defined by RQ-PCR for at least one leukemia-specific IG/TR gene rearrangement or leukemia specific genetic aberration with a sensitivity of at least 10-4) after induction treatment
Relapse free survival | two years
  Relapse free survival after two years
Molecular relapse | two years
  The proportion of patients with molecular relapse
Overall survival | two years
  Overall survival after two years
Death during induction | 42 days
  Death during induction
Death in complete remission | up to 2 years
  Death in complete remission

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Stelljes, MD, Principal Investigator — Universität Münster
Locations (14):
- Germany (14):
  - Klinikum Augsburg, Augsburg
  - Universität Bonn, Bonn
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Uniklinik Dresden, Dresden
  - University Hospital Düsseldorf, Düsseldorf
  - Universität Erlangen, Erlangen
  - Univeristätsklinikum Essen, Essen
  - University Hospital of Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Heidelberg
  - Uniklinikum, Jena
  - University of Muenster, Münster
  - Klinikum Nürnberg Nord, Nuremberg
  - Robert - Bosch - Krankenhaus, Stuttgart

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stelljes M, Raffel S, Alakel N, Wasch R, Kondakci M, Scholl S, Rank A, Hanel M, Spriewald B, Hanoun M, Martin S, Schwab K, Serve H, Reiser L, Knaden J, Pfeifer H, Marx J, Sauer T, Berdel WE, Lenz G, Bruggemann M, Gokbuget N, Wethmar K. Inotuzumab Ozogamicin as Induction Therapy for Patients Older Than 55 Years With Philadelphia Chromosome-Negative B-Precursor ALL. J Clin Oncol. 2024 Jan 20;42(3):273-282. doi: 10.1200/JCO.23.00546. Epub 2023 Oct 26. PMID 37883727